CLINICAL TRIAL: NCT01193686
Title: Evaluating a Peer Visitor Program for OIF/OEF Veterans With Polytrauma
Brief Title: Peer Visitation for OEF/OIF Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RRP 09-134
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Results first posted 2015-01-05 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-10

CONDITIONS: Polytrauma; Blast Injuries
MeSH Terms: conditions — Multiple Trauma; Blast Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peer Visitation Training (Peer Mentor) (Experimental): Veteran Peer Visitors participated in a 2-day training program and then provide at 1-5 visits to at least 2 recipients.
  Interventions: Other: Peer Visitation
- Peer Visitation (Experimental): Veterans who received at least one visit from a Veteran Peer Visitor.
  Interventions: Other: Peer Visitation

INTERVENTIONS:
Other: Peer Visitation — Trained Volunteers will visit OEF/OIF Veterans with Polytrauma Injuries to provide support.

SUMMARY:
The goal of this study was to train OIF/OIF Veterans with multiple injuries to be Peer Visitors, i.e., Volunteers who visit more recently OIF/OEF Veterans and provide support. We evaluated the effectiveness of the training, and any benefits that Volunteer Peer Visitors and the Recipients of Peer Visitors experienced as a result of participating in Peer Visitation.

DETAILED DESCRIPTION:
Peer visitation (PV) provides individuals newly dealing with a particular injury/ illness with an opportunity to interact with a peer who has successfully managed a similar condition. Interaction with a successful role model can provide credible social support and information, increase self-efficacy and teach coping strategies, which in turn can engender hope and motivation to engage in treatment and use active coping strategies. In spite of the widespread clinical availability of PV programs, the amount and type of training and clinical/organizational varies widely, and empirical support for their efficacy is limited. The main objective of this project is to test the feasibility of implementing a PV program for OEF/OIF veterans with war-related polytrauma.

The proposed study represented a unique opportunity to evaluate three important aspects of peer visitation among OEF/OIF Veterans. Our three hypotheses were: H 1: Veteran Peer Visitors (VPVs) who complete the training will demonstrate successful acquisition of efficacy, knowledge and skills as measured by: (1) pre- and post-tests administered before and after the training; (2) trainer evaluations upon completion of the training, (3) self-evaluation of at least two actual peer visits, and (4) evaluation by two individuals who receive peer visits. H2: VPVs who complete the study will demonstrate increased self-care, improved mood, and increased post-traumatic growth compared to pre-training baseline measures. H 3: Veterans who receive a visit from a VPV will endorse improvement in one or more of the following areas: stress, self-efficacy, activation, mood, ability to make meaning of their experiences, and knowledge of coping options.

We used a mixed-methods study to evaluate the feasibility of PV training materials developed in a previous grant to certify 12-18 Veteran Peer Visitors (VPVs). In a prior project, the proposed research team developed the training materials to be tested in this feasibility study, including screening tools to identify appropriate candidates for VPV training, an Instructor manual and a Veteran PV workbook.

Two types of participants: Veteran Peer Visitors and Recipients of VPVs were recruited via the Polytrauma Network Site in VISN 20 (Seattle). VPVs were nominated by a clinician to participate and, if enrolled, will undergo 2-day training and will be required to pass a test upon completion of training. Training included a VA Voluntary Services background check, and orientation to the VHA and VA privacy policies. VPVs became official VA volunteers. Each certified VPV was required to provide 1-5 visits to at least two Veterans. Both VPVs and recipients of VPV completed surveys at baseline and upon study completion.

ELIGIBILITY:
Inclusion Criteria:

For Peer Visitors:

* eligibility will be determined using a combination of self-assessment, clinician recommendation, and Voluntary Services screening

For participants who are interested in receiving a peer visitor:

* eligibility will be determined by the referring clinical team and the Research Nurse

Peer Visitors:

To be eligible to participate in the study as a potential Veteran Peer Visitor, Veterans must complete several screening steps. A Veteran must be nominated by a clinician from the Center for Polytrauma Care (CPC) Clinical Team, or they must nominate themselves for the project and seek endorsement from a clinician on the CPC team. To be nominated or endorsed by a clinician, the Veteran must have been observed by the clinical team member to demonstrate the following specific behaviors and characteristics:

* Reliable and organized about keeping appointments (80% adherence or better)
* Demonstrate excellent insight into own treatment goals, progress, barriers, treatment rationale
* Not demonstrate any "high-risk" behaviors in the previous 12 months, including suicidal ideation or intent, inpatient psychiatric treatment (other than planned, voluntary admission to Evaluation and Brief Treatment Unit), active substance abuse or dependence, uncontrolled psychotic symptoms (e.g., hallucinations, delusions), felonies.
* Evidence of good social support (i.e., clinician aware of supportive relationships)
* Engaged in meaningful life goals and activities (e.g., work, school, volunteering, parenting, recreation, church)
* Able to pass background check for Voluntary Services
* Must be English Speaking
* Able to complete pen and paper surveys

Exclusion Criteria:

* Not an OEF/OIF Veteran
* Under age 18
* Non English Speaking
* Psychiatrically at risk (i.e., uncontrolled psychotic symptoms, active substance abuse or dependence)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda M. Williams, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

REFERENCES:
- [Result] Williams RM, Bambara J, Turner AP. A scoping study of one-to-one peer mentorship interventions and recommendations for application with Veterans with postdeployment syndrome. J Head Trauma Rehabil. 2012 Jul-Aug;27(4):261-73. doi: 10.1097/HTR.0b013e3182585cb6. PMID 22767074

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Both types of study participants were recruited from Veterans who were seen in Polytrauma Clinics at the Polytrauma Network Site. Both types of participants were referred by clinicians based on their clinical knowledge of whether this intervention seemed indicated; Recipients could also self-refer based on printed information.
Pre-assignment Details: 400 Veterans were considered by the interdisciplinary polytrauma team as candidates for PV training. Of these, 29 (7%) were nominated. Of these, 14 (48%) were not enrolled: 6 (21%) due to time or travel restrictions, 6 (21%) could not be reached, and 2 (6%) because they had either been injured too recently or not participated in enough therapies.
Groups:
- Veteran Peer Visitors: Of the 15 (52%) PV who enrolled in the study and completed the baseline assessment, 4 (27%) withdrew prior to PV training due to moving out of state (3) or schedule limitations (n=1). One was removed from the study by investigators due to discovery of invalid reporting.
- Recipients of PV: 9 Veterans receiving care at a Polytrauma Network Site (of over 300 seen during the study period) expressed interest in meeting with a Veteran Peer Mentor. Of these 8 completed visits and all study requirements. One withdrew for non-study-related reasons.
Period: Overall Study
Arm/Group | Veteran Peer Visitors | Recipients of PV
Started | 15 | 9
Completed Baseline Assessment | 15 | 9
Completed Mentor Training | 9 | 0 (Not applicable. Recipients were not required to complete training.)
Completed Visits and Final Assessment | 8 | 8
Completed | 8 | 8
Not Completed | 7 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Removed by Investigators; unable to matc | 3 | 0

BASELINE CHARACTERISTICS:
Population: Descriptive demographics statistics were computed to characterize both baseline populations.
Groups:
- Veteran Peer Visitors: Veterans who seved in Operation Iraqi Freedom or Operation Enduring Freedom, sustained polytrauma injuries, and successfully completed rehabiliation were recruited for training as peer mentors.
- Recipients of Peer Visitors: Veterans who seved in Operation Iraqi Freedom or Operation Enduring Freedom, sustained polytrauma injuries, and were initiating rehabilitation therapies.
- Total: Total of all reporting groups
Arm/Group | Veteran Peer Visitors | Recipients of Peer Visitors | Total
Number analyzed (Participants) | 14 | 8 | 22
Age, Continuous [Mean (Full Range); unit: years] | 34.1 [26 to 62] | 36.5 [23 to 48] | 35 [23 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 13 | 7 | 20
Patient Health Questionnaire-9 [Mean (Full Range); unit: units on a scale] — The PHQ-9 assesses 9 symptoms of depression. Respondents are asked to indicate how often they have been bothered by each of the symptoms in the past two weeks, with response options ranging from 1 = "not at all" to 4 = "nearly every day". Possible total scores range from 9 (no symptoms of depression) to 36 (most severe depressive symptoms).
  units on a scale | 12 [9 to 15] | 27.4 [21 to 32] | 18.2 [9 to 32]
Self-Reported Anger [Mean (Full Range); unit: units on a scale] — This measure was developed for this study and included 5 items measuring "how angry you have felt in the last month". Sample items include: "I feel out of control with my anger" and "I'm so angry I feel like yelling or cursing at someone." Response options ranged from 1 = "strongly disagree" to 7 = "strongly agree". Possible total scores ranged from 5 to 35 with higher scores indicating greater feelings of anger.
  units on a scale | NA [NA to NA] — Not administered to Veteran Peer Visitors | 28.5 [17 to 35] | NA [NA to NA] — Only administered to Recipients of Peer Visitors
PTSD check-list (PCL) Military Version [Mean (Full Range); unit: units on a scale] — The PCL-M assesses the degree to which each of the 17 symptoms of PTSD outlined in the DSM-IV have been experienced in the past month. Possible response options range from 1 = "not at all" to 5 = "extremely". The scale also includes two questions that ask about the presence of traumatic events: "When the event(s) occurred, did you feel terrified?" and "When the event(s) occurred, did you feel helpless?", with the same response options. Total possible scores range from 19-95, with higher scores indicating greater PTSD symptomatology.
  units on a scale | 34 [21 to 46] | 68 [53 to 82] | 56 [21 to 82]
Patient Activation [Mean (Full Range); unit: units on a scale] — This measure was based on the Patient Activation Measure, and included 13 items reflecting self-efficacy for managing health/health care, active engagement in health care, and knowledge of health condition and treatment options. Possible scores ranged from 0-52, with higher scores indicating higher levels of efficacy, activation, and knowledge.
  units on a scale | NA [NA to NA] — This measure was not administered to Veteran Peer Visitors | 39 [14 to 43] | NA [NA to NA] — Only administered to Recipients of Peer VIsitors
Post Traumatic Growth Inventory [Mean (Full Range); unit: units on a scale] — This measure assesses emotional/psychological growth acquired by surviving a traumatic experience. Elements of post-traumatic growth can include increased sense of self, deepened relationships, appreciation for life, increased spirituality. Possible scores range from 0-105 with higher scores indicating more growth.
  units on a scale | 64.6 [23 to 98] | NA [NA to NA] — This measure was not administered to Recipients of Peer Visitors | NA [NA to NA] — Only administered to Veteran Peer Visitors

OUTCOME MEASURES:

1. Primary Outcome: Post Traumatic Growth Inventory
Description: Administered only to Peer Visitors, possible range 0-105, with higher scores indicating greater post-traumatic growth. Post-traumatic growth includes emotional changes such as noticing a stronger sense of self, deepened relationships, increased sense of gratitude or appreciation for life, increased spirituality.
Time Frame: Upon completion of study requirements (i.e., visits)
Population: This measure was only administered to Veteran Peer Visitors.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Veteran Peer Visitors | Recipients of PV
Number analyzed (Participants) | 8 | 0
units on a scale | 67.4 [21 to 90] |

2. Secondary Outcome: Patient Health Questionnaire-9 (Depression Screen)
Description: 9-item depression screen with possible response options ranging from 9-36, with higher numbers indicating greater depression symptom severity.
Time Frame: Upon completion of visits.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Veteran Peer Visitors | Recipients of PV
Number analyzed (Participants) | 8 | 9
units on a scale | 19.4 [13 to 30] | 23.6 [19 to 30]

3. Secondary Outcome: Post-Traumatic Stress Disorder Checklist- Military Version (PCL-M)
Description: Measures PTSD symptoms. Possible scores range from 19-95, with higher scores indicating greater symptom severity.
Time Frame: Upon study completion.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Veteran Peer Visitors | Recipients of PV
Number analyzed (Participants) | 8 | 9
units on a scale | 44.7 [23 to 76] | 53.7 [42 to 73]

4. Secondary Outcome: Patient Activation Measure
Description: Measures participante self-efficacy, knowledge of and engagement in health care. Possible scores range from 13-52 with higher scores indicating greater efficacy/knowledge/engagement.
Time Frame: Post- Participation
Population: This measure was only administered to Recipients of Peer Visitation.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Veteran Peer Visitors | Recipients of PV
Number analyzed (Participants) | 0 | 9
units on a scale |  | 38 [33 to 41]

5. Secondary Outcome: General Anger Level
Description: 5-item scale developed for this study. Assesses level of perceived experienced anger in the past month. Possible scores range from 5-35 with higher scores indicating greater levels of anger.
Time Frame: Post- Participation
Population: This measure was only administered to Recipients of Peer Visits.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Veteran Peer Visitors | Recipients of PV
Number analyzed (Participants) | 0 | 9
units on a scale |  | 24.8 [16 to 35]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Veteran Peer Visitors: Veteran Peer Visitors (VPV) who participated in a 2-day training program and then provided at 1-5 visits to at least 2 recipients. All Peer Visitors had served in Operation Iraqi Freedom or Operation Enduring Freedom, sustained polytrauma injuries, and successfully completed rehabilitation.
- Recipients of Veteran Peer Visitation: Veterans of Operation Enduring Freedom or Operation Iraqi Freedom who sustained polytrauma (i.e., mutiple systems involved) injuries.
Arm/Group | Veteran Peer Visitors | Recipients of Veteran Peer Visitation
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/9
Other Adverse Events (participants affected / at risk) | 0/15 | 0/9

LIMITATIONS AND CAVEATS:
We had great difficulty recruiting Recipients of Peer Visitors, i.e., Veterans who wished to receive mentorship from our trained peer visitors. This rendered our sample size too small for planned analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes